CLINICAL TRIAL: NCT01699412
Title: Randomized Double-blid Clinical Trial Comparing the Topical Treatment With Clobetasol and Dexamethasone for Oral Lesions of Chronic Graft-versus-host Disease in Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Clinical Trial With Clobetasol and Dexamethasone for Topical Treatment of Oral Lesions of Chronic Graft-versus-host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0712.1.146.000-08
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Graft vs Host Disease; Oral Manifestations
Keywords: Bone Marrow Transplantation; Graft vs Host Disease; Oral Manifestations
MeSH Terms: conditions — Graft vs Host Disease; Oral Manifestations | interventions — Clobetasol; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Patients under topical treatment with solution of dexamethasone 0.1 mg/mL associated to nystatin 100,000 UI/mL
  Interventions: Drug: Dexamethasone
- Clobetasol (Experimental): Patients under topical treatment with solution of clobetasol 0.05% associated with nystatin 100,000 UI/mL
  Interventions: Drug: Clobetasol

INTERVENTIONS:
Drug: Clobetasol — Rinse with a solution of clobetasol 0.05% associated to nystatin 100,000 UI/mL, for 1 minute, during 28 days
  Arms: Clobetasol
Drug: Dexamethasone — Rinse with a solution of dexamethasone 0.1 mg/mL associated to nystatin 100,000 UI/mL, for 1 minute, during 28 days
  Arms: Dexamethasone

SUMMARY:
The purpose of this study is to perform a randomized, double-blind, clinical trial comparing the topical treatment with clobetasol or dexamethasone for symptomatic oral lesions of chronic graft-versus-host disease.

DETAILED DESCRIPTION:
All patients with symptomatic oral lesions of cGVHD were included in the study. Exclusion criteria were patients with 12 years or less of age, history of allergy to any of the studied medications and patients already under other topical treatment for oral lesions of cGVHD. Patients were randomly assigned between two study groups: one group rinsed with a solution of clobetasol propionate 0.05% associated to nystatin 100,000 UI/mL; and another group rinsed with a solution of dexamethasone 0.1 mg/ml associated to nystatin 100,000 UI/mL. Patients were instructed to use the solution 3 times a day, during 1 minute, for 28 days. Clinical exams were performed at baseline and after 28 days. Patients were evaluated by an oral medicine expert, previously calibrated for evaluation of oral cGVHD lesions. Oral lesions of cGVHD were diagnosed according to NIH 2005 criteria, and graded according to the modified oral mucositis rating scale. Evaluation of the symptoms of the oral mucosa and of xerostomia were performed through visual analogue scale. Samples for fungal culture were obtained before and after the topical treatment. Results were submitted to a descriptive analysis. Chi-square was used for the comparison of categorical variables. Mann-Whitney and Wilcoxon tests were used for the comparison of measurable data inter and intra-groups, respectively. Significance level was set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic oral lesions of chronic graft-versus-host disease

Exclusion Criteria:

* Patients with less than 12 years of age
* Patients physically of mentally disabled
* History of allergy to any of the medications under study
* Patients already under topical treatment for oral lesions of chronic GVHD

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptoms related to oral cGVHD at 4 weeks | Baseline and 4 weeks
  Comparison of symptoms of oral lesions of chronic GVHD, analyzed through visual analogue scale, at baseline and after 4 weeks of topical treatment

SECONDARY OUTCOMES:
Change from baseline in clinical aspects of oral cGVHD at 4 weeks | Baseline and 4 weeks
  Comparison of the morphologic response of the oral lesions of chronic GVHD, measured through modified Oral Mucositis Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cesar W. Noce, DDS, MSD, Principal Investigator — Universidade Federal do Rio de Janeiro; Sandra R. Torres, DDS,MSD,PhD, Study Chair — Universidade Federal do Rio de Janeiro; Ângelo Maiolino, MD,MSD,PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (2):
- Brazil (2):
  - Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro
  - Hematology and Hemotherapy Center, Campinas, São Paulo

REFERENCES:
- [Background] Noce CW, Gomes A, Copello A, Barbosa RD, Sant'anna S, Moreira MC, Correa ME, Maiolino A, Torres SR. Oral involvement of chronic graft-versus-host disease in hematopoietic stem cell transplant recipients. Gen Dent. 2011 Nov-Dec;59(6):458-62; quiz 463-4. PMID 22313917